CLINICAL TRIAL: NCT04053751
Title: Effects of Open and Closed System Endotracheal Suctioning Methods on Suctioning Frequency and Amount of Secretion
Brief Title: Effects of Open and Closed System Suctioning on Suctioning Frequency and Amount of Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ilkin Yilmaz, Research Assisstant, Dokuz Eylul University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018.KB.SAG.025
Record Dates: First submitted 2019-08-09; First posted 2019-08-12 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Secretion; Excess, Salivation
Keywords: intensive care unit; endotracheal suctioning; open suctioning system; closed suctioning system; nursing
MeSH Terms: conditions — Sialorrhea

STUDY DESIGN:
Intervention Model Description: Randomized controlled crossover trial. There are two arms. open and closed suctioning systems (OSS vs CSS). the patients are randomized. They are monitorized for two days. If a patient is suctioned via OSS in the first enrolled day, the same patient is suctioned via CSS in the second enrolled day. For CSS, vice versa.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- closed suctioning system (Experimental): Closed suctioning system will be compared with open suctioning system
  Interventions: Procedure: closed suctioning system
- open suctioning system (No Intervention): The patient will be monitored with closed system for one day and open aspiration system on the other day.

INTERVENTIONS:
Procedure: closed suctioning system — a randomized allocated patient will be monitored for two days. Closed suctioning system will evaluate as experimental group. open suctioning system will evaluate as control group.
  Arms: closed suctioning system

SUMMARY:
Tracheal suctioning is a process which is often applied to patients' care who have an artificial airway and whose respiration is achieved via mechanical ventilation. When secretions are not cleaned enough, it causes a variety of complications in the patient from hypoxemia to infection.

It is reported that the studies with nurses in clinical practice have shown that they have opinions such as the closed system does not suction the patients effectively as the open system does; it remains incapable in removing secretions, thus the suctioning process is being applied more frequently.

Therefore this study is designed to examine the amount of secretions and frequency of suctioning as a result of open and closed suctioning systems.

DETAILED DESCRIPTION:
Patients will be monitored for two days. On the first day, the patient will be followed up with an open system and the second day closed suctioning system will be used, or the patient will be followed up with a closed system on the first day and followed with an open system on the second day. The patients are randomly allocated on the first follow up days. The follow-up period has two consecutive days. suctioning will be performed for 12 hours in one day. The number of suctions will be recorded. The amount of secretion will be accumulated in the mucus collection vessel. At the end of the day, the secretion will be weighed with precision weighing.

ELIGIBILITY:
Inclusion Criteria:

* orally intubated in first 96 hours
* stabilized patients in conditionally
* platelets > 50.000
* not have hemorrhagic secretions

Exclusion Criteria:

* hemodynamically unstabilized patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
frequency of suctioning | 12 hours of a day
  frequency of suctioning in a half of a day
amount of secretion | 12 hours of a day
  amount of secretion in a half of a day

SECONDARY OUTCOMES:
spo2 | 12 hours of a day
  differences in spo2 between open and closed suctioning systems
tidal volume | 12 hours of a day
  differences in tidal volume between open and closed suctioning systems

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Ozden, PhD, Study Director — Dokuz Eylul University Faculty of Nursing; Ilkin Yilmaz, PhD, Principal Investigator — Dokuz Eylul University Faculty of Nursing
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the patients data with other researchers.

REFERENCES:
- [Derived] Yilmaz I, Ozden D. The effects of open and closed system endotracheal suctioning methods on suctioning frequency, amount of secretion, and haemodynamics: A single-blind, randomised, 2 x 2 crossover trial. Aust Crit Care. 2024 Jan;37(1):25-33. doi: 10.1016/j.aucc.2023.09.002. Epub 2023 Oct 11. PMID 37833132